CLINICAL TRIAL: NCT00974025
Title: Vitamin C May Improve Endothelial Function and Exercise Capacity in Functional Single Ventricle Patients After Fontan Palliation
Brief Title: Impact of Vitamin C on Endothelial Function and Exercise Capacity in Fontan-Palliated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Griese-Hutchinson Champions for Children's Hearts Investigator Award (Unknown)
Responsible Party: Principal Investigator, John R. Charpie, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00029464
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Fontan Procedure; Hypoplastic Left Heart Syndrome; Tricuspid Atresia
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tricuspid Atresia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C (Experimental): High-dose Vitamin C in 4 age-based doses will be given in two-daily doses for four weeks
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Placebo will be given in two-daily doses for four weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — High-dose Vitamin C will be administered in 4 age-based dosing groups
  Arms: Vitamin C
Dietary Supplement: Placebo — Placebo will be administered twice daily for four weeks
  Arms: Placebo

SUMMARY:
In this study, investigators will evaluate the effect of vitamin C on endothelial function, exercise tolerance and quality of life in patients with a single ventricle who have been palliated to Fontan physiology. The hypothesis is that vitamin C will result in improved exercise tolerance and endothelial function in patients who have undergone the Fontan operation, compared to placebo.

DETAILED DESCRIPTION:
Recent evidence suggests that after Fontan operation, single ventricle patients have impaired function of the vascular endothelium due in part to abnormalities in nitric oxide signaling. Endothelial dysfunction may contribute to the development of congestive heart failure and exercise intolerance that have been well-documented in Fontan patients. Therapeutic interventions to improve endothelial function in adults with heart failure have mainly focused on increasing the synthesis or decreasing the degradation of nitric oxide. We propose a randomized, prospective, placebo-controlled trial of vitamin C, an antioxidant that protects NO deactivation, in subjects with single ventricular anatomy after Fontan palliation. The specific aims of this study are to compare NO signaling, endothelial function and exercise capacity in Fontan subjects to that of a control group that is frequency-matched to case subjects by age and sex, and to assess NO signaling, endothelial function and exercise capacity in Fontan subjects after 4 weeks of oral vitamin C (or placebo) therapy. These results have particular importance because improving the endothelial response in Fontan patients has the potential to reduce the risk of developing congestive heart failure and improve exercise capacity. Furthermore, assessing endothelial function and the effects of therapies aimed at improving vascular health may be generalizable to many other chronic pediatric conditions associated with increased cardiovascular risk such as obesity, diabetes mellitus, and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 8-25 years of age
* Fontan-palliated patient

Exclusion Criteria:

* New York Heart Association (NYHA) classes III or IV
* Diabetes mellitus
* Family history of premature coronary artery disease
* Use of Sildenafil or other pulmonary artery vasodilators
* Prior cardiac arrest (outside the first 24-hours postoperatively)
* Life-threatening dysrhythmias
* Severe ventricular dysfunction
* Severe AV valve regurgitation
* Pregnancy
* Severe renal or hepatic impairment

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption (from baseline to post-study drug testing) | 4 weeks

SECONDARY OUTCOMES:
Oxygen Pulse | 4 weeks
Peak Work | 4 weeks
Endo-PAT score | 4 weeks
Framingham Modified Endothelial Function Score | 4 weeks
PedsQL 4.0 - quality of life assessment | 4 weeks
BNP | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John R Charpie, MD, Study Director — University of Michigan; Bryan H Goldstein, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Goldstein BH, Golbus JR, Sandelin AM, Warnke N, Gooding L, King KK, Donohue JE, Gurney JG, Goldberg CS, Rocchini AP, Charpie JR. Usefulness of peripheral vascular function to predict functional health status in patients with Fontan circulation. Am J Cardiol. 2011 Aug 1;108(3):428-34. doi: 10.1016/j.amjcard.2011.03.064. Epub 2011 May 19. PMID 21600541
- [Derived] Goldstein BH, Sandelin AM, Golbus JR, Warnke N, Gooding L, King KK, Donohue JE, Yu S, Gurney JG, Goldberg CS, Rocchini AP, Charpie JR. Impact of vitamin C on endothelial function and exercise capacity in patients with a Fontan circulation. Congenit Heart Dis. 2012 May-Jun;7(3):226-34. doi: 10.1111/j.1747-0803.2011.00605.x. Epub 2011 Dec 18. PMID 22176653